CLINICAL TRIAL: NCT01484340
Title: A Smoking Cessation Trial in HIV-infected Patients in South Africa
Acronym: JHU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Witwatersrand, South Africa (Other); Truth Initiative (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00048461; 1R01DA030276-01A1 (NIH)
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Results first posted 2018-11-06 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Smoking Cessation; HIV
Keywords: smoking; administration, cutaneous
MeSH Terms: conditions — Smoking Cessation; Smoking | interventions — Nicotine; Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Counseling only (Experimental): Participants in this arm will receive advice to quit smoking and self-help materials from the study interventionist in a standardized fashion (intensive anti-smoking counseling).
  Interventions: Behavioral: Intensive Counseling
- Nicotine Replacement Therapy +counseling (Experimental): Participants in this arm will receive the nicotine patch in addition to the intensive anti-smoking counseling. Participants will receive instruction on proper use of the nicotine patch (i.e., placement, use of one patch a day, importance of not smoking while using the patch, and tapering of patches).
  Interventions: Drug: Nicotine; Behavioral: Intensive Counseling

INTERVENTIONS:
Drug: Nicotine — The nicotine patch be given in three phases:
  * 2 weeks of patches at enrollment
  * 6 weeks of patches at two-week follow-up visit
  * 2 weeks of patches at two-month follow-up visit
  This schedule will cover the entire 10-week course of therapy as per label instructions: 6 weeks at 21mg; 2 weeks at 14mg; and 2 weeks at 7mg.
  Other Names: Nicorette
  Arms: Nicotine Replacement Therapy +counseling
Behavioral: Intensive Counseling — The advice to quit smoking message will follow NCI's 5A's model for smoking cessation counseling. This is a simple smoking cessation counseling strategy with 5 discrete components: (1) Ask about smoking at every opportunity; (2) Advise the patient to quit smoking; (3) Assess readiness to quit; (4) Assist the patient in quitting; and (5) Arrange follow-up.
  Visit schedule:
  * Baseline
  * 2-week follow-up (Quit Day)
  * 1-month follow-up
  * 2-month follow-up
  * 3-month follow-up
  * 6-month follow-up
  Participants abstinent at 6-month follow-up will be next seen at 12-month follow-up.
  Participants still smoking at 6-month follow-up will be offered group-assigned intervention again.

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial (RCT) of intensive anti-smoking counseling plus nicotine replacement therapy versus intensive anti-smoking counseling alone among HIV-infected patients in South Africa, and to concurrently measure the prevalence of smoking among HIV-infected patients in South Africa.

DETAILED DESCRIPTION:
Tobacco use is estimated to be responsible for over 5 million deaths globally every year and HIV/AIDS kills 2 million worldwide, with persons living in the developing world especially at risk. However, the association between tobacco use and HIV is not clearly understood. The introduction of highly active antiretroviral therapy (HAART) has led to longer duration of survival following HIV-infection in the developed world, and now that HAART is being rolled out in the developing world, survival will increase in these highly endemic regions as well. Given this increase in survival, more people will die of non-HIV related illnesses for which smoking plays an important causal role. Smoking cessation for HIV-infected persons has been studied in the US though these studies have had small numbers and limited follow-up. US based studies suggest that approaches that combine nicotine replacement therapy (NRT) and counseling interventions are most successful. Optimal approaches in resource-limited settings have not been determined.

This study will compare intensive counseling plus NRT versus intensive counseling only, comparing smoking cessation at 2, 6 and 12 months. At 6 months, patients who are still current smokers will be given a second opportunity to receive their group assigned intervention, either intensive counseling plus NRT or intensive counseling alone. We will relate smoking exposure and cessation to HIV progression as measured by immunologic and viral markers, risk of respiratory infections, including tuberculosis, and AIDS-related malignancies. The RCT will be performed at the Tshepong HIV Wellness Clinic in Klerksdorp, South Africa, associated with the Reproductive Health & HIV Research Unit of the University of the Witwatersrand, South Africa.

ELIGIBILITY:
Inclusion Criteria:

* Current, daily smoker (biochemically verified via a positive result on the SmokeScreen® test from GFC Diagnostics Ltd., as described in the outcomes)
* Be willing to set a quit date within 2 weeks after baseline assessment
* Agree to participate in study and anticipated to be attending Tshepong Wellness Clinic, Jouberton Community Health Center, or Grace Mokhomo Community Health Center (due to HIV infection) for at least 6 months

Exclusion Criteria:

* Pregnant or nursing
* Currently using smokeless tobacco (including electronic cigarettes, NRT or other cessation treatment)
* Tuberculosis confirmed case
* Weight <45 kg or BMI <20
* Suffering from any unstable medical condition which could preclude use of the nicotine patch:

  * unstable angina
  * uncontrolled hypertension
  * active skin disease (e.g. psoriasis)
  * history of skin allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Golub, PhD, Principal Investigator — Johns Hopkins University
Locations (3):
- South Africa (3):
  - Grace Mokhomo Community Health Center, Klerksdorp, North West
  - Jouberton Community Health Center, Klerksdorp, North West
  - Tshepong Wellness Clinic, Klerksdorp, North West

REFERENCES:
- See also: 5 As: Treating Tobacco Use and Dependence — http://www.ahrq.gov/clinic/tobacco/5steps.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Counseling Only: Participants in this arm will receive advice to quit smoking and self-help materials from the study interventionist in a standardized fashion (intensive anti-smoking counseling).
  Intensive Counseling: The advice to quit smoking message will follow NCI's 5A's model for smoking cessation counseling. This is a simple smoking cessation counseling strategy with 5 discrete components: (1) Ask about smoking at every opportunity; (2) Advise the patient to quit smoking; (3) Assess readiness to quit; (4) Assist the patient in quitting; and (5) Arrange follow-up.
  Participants abstinent at 6-month follow-up will be next seen at 12-month follow-up.
  Participants still smoking at 6-month follow-up will be offered group-assigned intervention again.
- Nicotine Replacement Therapy +Counseling: Participants in this arm will receive the nicotine patch in addition to the intensive anti-smoking counseling. Participants will receive instruction on proper use of the nicotine patch (i.e., placement, use of one patch a day, importance of not smoking while using the patch, and tapering of patches).
  Nicotine: The nicotine patch be given in three phases:
  * 2 weeks of patches at enrollment
  * 6 weeks of patches at two-week follow-up visit
  * 2 weeks of patches at two-month follow-up visit
  Intensive Counseling: same as in "Counseling only" arm
  Participants abstinent at 6-month follow-up will be next seen at 12-month follow-up.
  Participants still smoking at 6-month follow-up will be offered group-assigned intervention again.
Period: Overall Study
Arm/Group | Counseling Only | Nicotine Replacement Therapy +Counseling
Started | 281 | 279
Completed | 281 | 279
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Counseling Only | Nicotine Replacement Therapy +Counseling | Total
Number analyzed (Participants) | 281 | 279 | 560
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 36 [30 to 44] | 39 [32 to 46] | 37 [31 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 55 | 123
  Male | 213 | 224 | 437
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African/Black | 281 | 276 | 557
  Race: Colored | 0 | 1 | 1
  Race: Indian/Asian | 0 | 1 | 1
  Race: Not documented | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  South Africa | 281 | 279 | 560
Number of cigarettes smoked per day [Median (Inter-Quartile Range); unit: cigarettes per day] | 10 [6 to 15] | 9 [5 to 15] | 10 [5 to 15]

OUTCOME MEASURES:

1. Primary Outcome: Smoking Status Using a Point of Care Test for Measuring Carbon Monoxide (CO)
Description: A point of care test for measuring carbon monoxide (CO) will be conducted via the piCO Smokerlyzer from OPS Medical, designed specifically for smoking cessation programs and tobacco control programs. Carbon monoxide will be measured in an exhaled breath in parts-per-million (ppm). A reading of ≤ 7ppm will indicate abstinence.
Time Frame: 6 months from baseline
Population: As treated analysis: Patients without biochemical verification at any visit were excluded from the denominator. Counseling only arm: 53 patients excluded. Nicotine Replacement Therapy +counseling arm: 54 patients excluded.
Measure: Median (Inter-Quartile Range); unit: COppm
Arm/Group | Counseling Only | Nicotine Replacement Therapy +Counseling
Number analyzed (Participants) | 228 | 225
COppm | 11 [5 to 19] | 11 [6 to 18]

2. Primary Outcome: Smoking Status Using a Point of Care Test for Measuring Cotinine
Description: A point of care urine test for measuring cotinine will also be conducted via the SmokeScreen® test from GFC Diagnostics Ltd. to verify smoking status. A reading of < 0.4 μg/ml cotinine equivalent will indicate abstinence.
Time Frame: 6 months from baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: μg/ml cotinine equivalent
Arm/Group | Counseling Only | Nicotine Replacement Therapy +Counseling
Number analyzed (Participants) | 228 | 225
μg/ml cotinine equivalent | 1.7 [0.5 to 4.7] | 1.5 [0.3 to 5.3]

3. Secondary Outcome: Smoking Status (COppm)
Description: A point of care test for measuring CO will be conducted via the piCO Smokerlyzer from OPS Medical, designed specifically for smoking cessation programs and tobacco control programs. Carbon monoxide will be measured in an exhaled breath in parts-per-million (ppm). A reading of ≤ 7ppm will indicate abstinence.
Time Frame: 2 months from baseline
Population: As treated analysis: Patients without biochemical verification at any visit were excluded from the denominator. Counseling only arm: 64 patients excluded. Nicotine Replacement Therapy +counseling arm: 60 patients excluded.
Measure: Median (Inter-Quartile Range); unit: COppm
Arm/Group | Counseling Only | Nicotine Replacement Therapy +Counseling
Number analyzed (Participants) | 217 | 219
COppm | 9 [4 to 17] | 11 [5 to 18]

4. Secondary Outcome: Smoking Status (COppm)
Description: as for outcome 3
Time Frame: 12 months from baseline
Population: As treated analysis: Patients without biochemical verification at any visit were excluded from the denominator. Counseling only arm: 72 patients excluded. Nicotine Replacement Therapy +counseling arm: 74 patients excluded.
Measure: Median (Inter-Quartile Range); unit: COppm
Arm/Group | Counseling Only | Nicotine Replacement Therapy +Counseling
Number analyzed (Participants) | 209 | 205
COppm | 10 [5 to 17] | 10 [5 to 17]

ADVERSE EVENTS:
Arm/Group | Counseling Only | Nicotine Replacement Therapy +Counseling
All-Cause Mortality (participants affected / at risk) | 3/281 | 4/279
Serious Adverse Events (participants affected / at risk) | 4/281 | 5/279
Other Adverse Events (participants affected / at risk) | 0/281 | 0/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Counseling Only (N=281) | Nicotine Replacement Therapy +Counseling (N=279)
Acute renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Tuberculosis (Infections and infestations) | 1 (1) | 2 (2) — Disseminated TB
Hospitalization (General disorders) | 1 (1) | 1 (1)
Lymphoma (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Age with dehydration (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No